CLINICAL TRIAL: NCT07260136
Title: A Study of Cervical Spine Abnormalities Associated With Down Syndrome in Children at Sohag University
Brief Title: Cervical Spine Abnormalities in Down Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, EsraaAMahmoud, Resident physician in pediatric department at sohag university, Sohag University
Other Study IDs: Soh-Med-25-7_17MS
Record Dates: First submitted 2025-09-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome; Cervical Spine Instability in Down Syndrome
Keywords: Cervical abnormalities associated with Down syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to determine the prevalence,clinical presentations and radiographic cervical spine abnormalities associated Down syndrome in children at sohag university hospital

ELIGIBILITY:
Inclusion Criteria:

* All patients attending to pediatric inpatient and outpatient clinics aged from 2y up to 18 y

Exclusion Criteria:

* children with other clinical syndromes Children with other neurological disorders (eg. Cerebral palsy , myopathy, neuropathy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Aims to study the prevalence, clinical presentationsand radiographic cervical spine abnormalities associated with Down syndrome in children at sohag university hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence, clinical presentations and radiographic cervical spine abnormalities associated with Down syndrome through study completion an average of 1 year . | Asses the perivlance of cervical spine abnormalities in patient with Down syndrome of patients aged from 2 years up to 18 years ,using measure tool atlanoaxial instability in ct neck (ADI>3ml)and other mutliple measures ex(weight,height,eg.)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No